CLINICAL TRIAL: NCT02177591
Title: Observational Study of the Association Between Periodontal Disease and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L14-141
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Periodontal Disease; Coronary Artery Disease
MeSH Terms: conditions — Periodontal Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CAD and MI: Patients with a history of coronary artery disease who have had a myocardial infarction in the past.
- CAD, no MI: Patients who have a history of coronary artery disease and have not had a myocardial infarction in the past.
- no CAD: Patients with no documented history of coronary artery disease.

SUMMARY:
The prevalence of cardiovascular disease is rising; new methods must be created to assess the cardiovascular status of patients. If cardiovascular disease can be predicted, it may facilitate prevention. An association between periodontal disease and cardiovascular has been established, but a definitive mechanism is not understood. A good first step in finding that mechanism is to look at the correlation between periodontal disease and cardiovascular disease, both of which have an inflammatory component. This study observes the level of cardiovascular disease in patients and correlates it with the presence and degree of periodontal pathogens.

DETAILED DESCRIPTION:
A possible association between periodontal disease and cardiovascular disease was first hypothesized in the 1980s. Epidemiological studies performed over the last 20 years have shown a strong correlation between periodontal disease and cardiovascular disease. However, the literature is somewhat divided, as some studies have shown moderate correlation while others have shown independent (insignificant) correlations between the two. This leaves a gap in the investigators knowledge that must be brought together through specific studies. There have been reports made to suggest that 52% of atherosclerotic plaques studied have been found to contain the same pathogens that cause periodontitis. This is the reason that these are the bacteria that will be focused on during the course of this study.

Periodontal disease, known as either gingivitis or periodontitis, is caused by the presence of bacteria in the gingival pockets in the mouth which over time can cause systemic inflammation through endotoxin production. Some examples of the bacteria that cause periodontal disease include Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans. These are gram-negative, anaerobic bacteria that are able to thrive in the sub-gingival space after they are able to successfully become established. These two bacteria have been known to invade oral epithelial cells, creating the possibility that they could invade epithelial cells elsewhere such as in coronary vessels. These bacteria will be cultured from the patient and the relative amounts of them as determined by culture techniques will be used to assess the prevalence of periodontal disease in the patient. P. gingivalis is of special importance because it is known to be found in patients with active periodontal disease and not commonly found in patients without periodontal disease. It can be identified by the black pigment produced upon culture. Tryptic Soy-Serum-Bacitracin-Vancomycin (TSBV) Agar is a selective medium that is able to isolate A. actinomycetemcomitans. The identity of A. actinomycetemcomitans can be confirmed based on the growth of "star-like" colonies on the TSBV Agar that are catalase positive. The relative amount of these bacteria as determined by culture will be used to correlate with the level of coronary artery disease based on the groups that each subject is assigned to. This is how the basis for an association between the two conditions can be determined.

Systemic inflammation occurs as a result of the release of pro-inflammatory cytokines in response to an infection. Some of the cytokines released, include high sensitivity C-reactive protein (hs-CRP), interleukin-1 (IL-1), and interleukin-6 (IL-6). Hs-CRP is a protein that is active during the acute phase response to inflammation. Its level in the blood has been shown to be markedly raised in chronic inflammation and has consistently been found to be elevated in patients with acute coronary syndromes. IL-1 is a pro-inflammatory cytokine that is also released as a result of systemic inflammation. Specifically, it has been found to be secreted in response to lipopolysaccharide (LPS) from gram-negative bacteria and has been found to be elevated in patients with increased periodontal disease. IL-6, like IL-1, is a pro-inflammatory cytokine that is part of the acute phase response to infection. It has been strongly correlated with increasing levels of coronary artery disease and has even been demonstrated as a predictive marker of mortality in Coronary Artery Disease (CAD). In addition to its role in CAD, IL-6 has also been found to be elevated in periodontal disease, creating the possibility for the basis of the link between these two diseases.

The aim of this study is to achieve a better understanding of the relationship between periodontal disease and coronary artery disease by correlating the severity of coronary artery disease with the presence and amount of the periodontal pathogens P. gingivalis and A. actinomycetemcomitans. The level of systemic inflammation caused by these pathogens and and coronary artery disease will also be assessed. This will determine if coronary artery disease can be associated with one of these specific pathogens more than the other and what levels of systemic inflammation can be associated with both of these conditions together.

Samples will be obtained from periodontal tissue, cultured, and the amount of the specified pathogens present will be correlated with the type and extent of the patient's cardiovascular disease. Blood tests will also be taken to assess the level of systemic inflammation occurring as a result of periodontal disease and cardiovascular disease.

Subjects will be assigned to one of 3 groups based on their cardiovascular status:

* Group 1 will include patients with no known history of CAD.
* Group 2 will include patients with a known history of CAD without previous Myocardial Infarction (MI).
* Group 3 will include patients with a known history of CAD and previous MI.

Charts for patients to be seen in the Cardiology clinic will be pre-screened by a member of the study team to determine if the patient is eligible for the study. Patients will be consented in a private setting and a cardiovascular disease history pertinent to the study will be taken for each patient who consents to participating in the study. Clean floss that has been will be used to collect a sample of gingival fluid from between the lower teeth of the patient. No measures have been taken to sterilize the floss, so appropriate aseptic techniques including the use of sterile gloves to prevent cross contamination. Three samples will be collected: in the midline of the teeth, behind the right or left lateral incisor, and in front of the right or left first molar. The decision to sample the right or left of the patient's mouth will be randomized (coin flip) unless the patient is missing teeth on one side and the sample must be taken from the side that will yield a proper sample. At least 2 out of the 3 samples must be obtained. These samples will be placed in 3 labeled (by study identification number and site of sample) sealed vials of thioglycollate broth and cultured for 48 hours. A sample will then be removed from the bottom of thioglycollate medium using a pipette (to extract anaerobic bacteria) and cultured on specific media for the presence of P. gingivalis, and A. actinomycetemcomitans using anaerobic precautions in the University Medical Center (UMC) microbiology laboratory. P. gingivalis will be cultured on a specialized Columbia agar supplemented with sheep's blood, bacitracin, colistin, and nalidixic acid to select for the isolation of P. gingivalis. A. actinomycetemcomitans can be isolated using a specialized tryptic soy-serum-bacitracin-vancomycin (TSBV) agar, a specialized agar that inhibits gram-positive and gram-negative aerobes and anaerobes. Each sample will be streaked onto an agar plate that has been labeled with the study ID and tooth location. The bacteria will be cultured using the quad-streak method and cultured for 24-48 hours and the pathogenic bacteria will be identified. P. gingivalis will be identified based on the growth of black pigmented colonies on the selective agar and A. actinomycetemcomitans will be identified based on the growth of star-like colonies on the TSBV agar. The level of periodontal disease in the patient will be assessed by the amount of growth on the plates, with a number assigned to each quadrant that the bacteria grow in. if they only grow in the first quadrant, they will be given a number designation of 1, and growth in the second through fourth quadrants will be designated by 2 through 4 respectively. Using this method, the level of the bacteria can be quantified, with 4 being the designation for highest relative amount of bacteria. The level of each pathogen found in the patients' mouths will be correlated with the severity of coronary artery disease in order to determine if there is a significant correlation. It will also be determined if one of the pathogens can be correlated with the severity.

In addition to the gingival sampling, a small portion (3 mL or 0.6 tsp) of the patient's blood will be used to test for hs-CRP, IL-6, and IL-1 as systemic markers of inflammation. The sample used will be taken during the initial clinic visit when the patient has given consent and the gingival sample is taken. The sample will be drawn by a nurse in order to obtain the necessary tests. 1 mL (0.2 tsp) of serum will be drawn for each test (0.6 tsp total) and sent to the UMC pathology lab for analysis. These levels will be compared to the normal values of IL-1 (0-5 pg/mL) and IL-6 (5-15 pg/mL) while hs-CRP will be correlated based on increasing levels. This will allow determination of the level of systemic infection caused by periodontitis (based on IL-1 level), coronary artery disease (based on hs-CRP level), or both (based on IL-6 level). Individual results will be recorded for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known CAD with and without previous MI, OR
* Patients with no known CAD
* Ages 18-89 years

Exclusion Criteria:

* Patients with a known history of rheumatoid arthritis.
* Patients with a known history of lupus.
* Patients currently under the care of a rheumatologist.
* Patients who have had a MI in the two weeks prior to entering the study.
* Patients with a previous history of coronary artery bypass graft.
* Patients who have taken antibiotics in the two weeks prior to entering the study.
* Patients who are unable to provide at least 2 out of the 3 gingival samples.
* Current smokers.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients from ages 18-89 years who are being seen in the Cardiology clinic at TTUHSC who meet inclusion and exclusion criteria, and who will consent to participating in the study. There will be 20 to 30 patients in each group.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparing level of coronary artery disease with amount of bacteria in the mouth | Baseline
  Will compare patients in each group with the numerical value of P. gingivalis and A. actinomycetemcomitans in the mouth.
Compare level of hs-CRP with level of bacteria | Baseline
  Will compare levels of hs-CRP (mg/dL) in the blood with the numerical value of P. gingivalis and A. actinomycetemcomitans in the mouth.
Compare levels of IL-6 with level of bacteria | Baseline
  Will compare levels of IL-6 (pg/mL) in the blood with the numerical value of P. gingivalis and A. actinomycetemcomitans in the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shurmur, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No